CLINICAL TRIAL: NCT00575224
Title: Pegasys and Copegus for Asian Patients With Treatment-naive Hepatitis C Genotypes 6, 7, 8, 9: a Phase IV, Randomized, Open-labeled, Multicenter Trial Comparing 24-week vs. 48-week Therapy
Brief Title: Pegasys and Copegus for Asian Patients With Treatment-naive Hepatitis C Genotypes 6, 7, 8, 9
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacific Health Foundation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Pacific Health Foundation: Mindie Nguyen, MD, MAS and Huy Trinh, M.D., Pacific Health Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEG-183; IRB Protocol #20041038; IRB Study #1059635
Record Dates: First submitted 2007-12-15; First posted 2007-12-18 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Hepatitis C; Asian Americans; Novel Genotypes; Treatment
Keywords: Hepatitis C; Genotype 6; Novel genoytpe; HCV; Treatment
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Pegylated interferon and ribavirin for 24 weeks
  Interventions: Drug: Pegylated interferon and ribavirin
- B (Other): Pegylated interferon and ribavirin for 48 weeks
  Interventions: Drug: Pegylated interferon and ribavirin

INTERVENTIONS:
Drug: Pegylated interferon and ribavirin — 180 ug of peg-IFN per week and 1000-1200 mg of ribavirin per day (weight-dependent). Treatment duration is determined by treatment arm.
  Other Names: Pegasys and Copegus

SUMMARY:
The purpose of this research study is to test the safety, tolerability, and effectiveness of the drugs Pegasys and Copegus when used for hepatitis C genotypes 6, 7, 8, and 9. Patients are randomly assigned (by chance) to either Treatment Group A (Pegasys and Copegus for 24 weeks) or Treatment Group B (Pegasys and Copegus for 48 weeks).

ELIGIBILITY:
Inclusion Criteria:

The subject must meet the following criteria for entry.

* Subject must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Adult subjects 18-70 years of age of both gender and any race as long as they have HCV genotype 6, 7, 8, and 9.
* Serum positive for HCV-RNA by PCR (qPCR) assay, or bDNA
* Liver biopsy within 24 months prior to entry to this protocol with a pathology report confirming that the histological diagnosis is consistent with chronic hepatitis C with stage II or more fibrosis. Biopsy must be scored or be re-read to score fibrosis stage and grade and severity of steatosis.
* Compensated liver disease with the following minimum hematologic, biochemical, and serologic criteria at the Entry Visit (WNL = within normal limits).

  * Hemoglobin (Hb) greater than or equal to12 gm/dL for women and 13 gm/dL for men.
  * White blood cell count (WBC) greater than or equal to 2,000/mm3
  * Platelets (PLT) greater than or equal to 90,000/mm3
  * Direct bilirubin (DB) less than or equal to 1.0
  * Indirect bilirubin (IB) = WNL or greater than or equal to 3.0 mg/dL if this is due to non-hepatitis related factors such as Gilbert's disease.
  * Creatinine (Cr) clearance greater than or equal to50 mL/minute or serum Cr greater than or equal to 1.5x UNL at screening.
* Fasting glucose (FBS) less than or equal to160 mg/dL and Hb A1c greater than or equal to 8.5% for diabetic subjects (whether on medication or diet controlled).
* Thyroid Stimulating Hormone (TSH) = WNL (Subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met.)
* Serum anti-HIV = negative
* Serum HBsAg = negative
* Abdominal ultrasound negative for liver masses within 3 months prior to entry. Patients without cirrhosis or transition to cirrhosis may have there imaging studies done within 12 months of study entry.
* Alpha-fetoprotein (AFP) less than or equal to 20 ng/mL obtained within 3 months prior to entry. Patients with 20 ng/mL less than or equal to AFP less than or equal to 100ng/mL may be enrolled after a normal biphasic abdominal CT within the previous 3 months if patients have Stage III/IV fibrosis and after a normal ultrasound if patients have Stage I/II fibrosis. If AFP is more than 100 but less than 200 ng/dL, all patients need to have a negative biphasic CT within 3 months.
* Female subjects must not be breast-feeding.
* A pregnancy test must be obtained within 24 hours to the first dose of study drugs and must be negative.
* Additionally, all fertile males and females must use two reliable forms of effective contraception (combined) during treatment with study drugs and 6 months after treatment completion.
* Acceptable forms of contraception may include intrauterine device, oral contraceptives, progesterone implanted rods [Norplant], medroxyprogesterone acetate [Depo-Provera], surgical sterilization, barrier method [diaphragm + spermicide or condom + spermicide]

Exclusion Criteria:

The subject will be excluded from entry if any of the following criteria apply:

* Women who are pregnant or breast feeding.
* Male partners of women who are pregnant.
* Suspected hypersensitivity to interferon, PEG-interferon or Copegus.
* Treatment with any investigational drug within 45 days of entry to this protocol.
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment greater than or equal to6 months prior to the first dose of study drug, except PEG-IFN alfa-2b and ribavirin. This includes amantadine, mycophenolate mofetil, thymosine alpha, viramidine, levovirin, supraphysiologic doses of steroids (greater than or equal to 10 mg/d for greater than or equal to 14 consecutive days of prednisone or equivalence) and radiation, exception: patients who have had a limited (greater than or equal to 7 day) course of acyclovir or valacyclovir for herpetic lesions more than 1 month prior to the first administration of test drug are not excluded.
* Any other cause for the liver disease other than chronic hepatitis C including but not limited to:

  * Co-infection with HBV
  * Hemochromatosis (iron deposition greater than or equal to2+ or severe in liver parenchyma)
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Significant obesity-induced liver disease (elevated ALT with BMI greater than or equal to 30)
  * Drug-related liver disease
* Hemophilia or any other condition that would prevent the subject from having a liver biopsy, including anticoagulant therapy.
* Hemoglobinopathies (e.g., Thalassemia) with significant anemia.
* History or other evidence of decompensated liver disease or a Child-Pugh score 6. Coagulopathy, hyperbilirubinemia, hepatic encephalopathy, hypoalbuminemia, ascites, and bleeding from esophageal varices are conditions consistent with decompensated liver disease.
* Patients with history of hepatocellular carcinoma.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the protocol such as:

  * A history of preexisting psychiatric condition, especially severe depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt are excluded. Severe depression would include the following: (a) subjects who have been hospitalized for depression, (b) subjects who have received electroconvulsive therapy for depression, or (c) subjects whose depression has resulted in a prolonged absence of work and/or significant disruption of daily functions. Subjects with a history of mild depression may be considered for entry into the protocol provided that a pretreatment assessment of the subject's mental status supports that the subject is clinically stable. The Investigator will formulate a management plan for each of the subjects that will become a part of the subject's medical record. The management plans may be developed in conjunction with a health care professional trained in psychology. For these subjects, the Investigator will review the subject's mental status at every visit.
  * CNS trauma or active seizure disorders requiring medication.
  * Significant cardiovascular dysfunction within the past 12 months (e.g., angina, congestive heart failure, recent myocardial infarction, severe uncontrolled hypertension or significant arrhythmia). Subjects with ECG showing clinically significant abnormalities.
  * Poorly controlled diabetes mellitus.
  * Chronic pulmonary disease (e.g., chronic obstructive pulmonary disease), documented pulmonary hypertension.
  * Immunologically mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], rheumatoid arthritis, idiopathic thrombocytopenia purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, clinical cryoglobulinemia with vasculitis).
  * Clinical gout.
  * Any patient with an increased baseline risk for anemia (e.g. thalassemia other than thalassemia trait, spherocytosis, history of GI bleeding, etc) or for whom anemia would be medically problematic
  * Patients in whom, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (40 g/L) (as may be seen with ribavirin therapy) would not be well-tolerated.
  * History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis etc.)
  * History of major organ transplantation with an existing functional graft
* Substance abuse, such as alcohol (greater than or equal to 80 gm/day), IV drugs and inhaled drugs. If the subject has a history of substance abuse, to be considered for inclusion into the protocol, the subject must have abstained from using the abused substance for at least 12 months. Stable subjects enrolled in a methadone maintenance program for at least one year may be enrolled if they are otherwise eligible and are monitored throughout the study for illicit drug use.
* Subjects not willing to abstain from the consumption of alcohol.
* Subjects with severe retinopathy (e.g. CMV retinitis, macular degeneration) or clinically significant retinal abnormalities.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.
* Any other condition, which in the opinion of the Investigators would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response | 24 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mindie H Nguyen, M.D., M.A.S., Principal Investigator — Stanford University Medical Center and Pacific Health Foundation
Locations (5):
- United States (5):
  - San Diego Gastroenterology Clinic, San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Westminster Gastroenterology Clinic, Westminster, California
  - Houston Gastroenterology Clinic, Houston, Texas
  - Digestive Health Associates of Texas, Plano, Texas

REFERENCES:
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] Adams NJ, Chamberlain RW, Taylor LA, Davidson F, Lin CK, Elliott RM, Simmonds P. Complete coding sequence of hepatitis C virus genotype 6a. Biochem Biophys Res Commun. 1997 May 19;234(2):393-6. doi: 10.1006/bbrc.1997.6627. PMID 9177282
- [Background] Nguyen MH, Keeffe EB. Prevalence and treatment of hepatitis C virus genotypes 4, 5, and 6. Clin Gastroenterol Hepatol. 2005 Oct;3(10 Suppl 2):S97-S101. doi: 10.1016/s1542-3565(05)00711-1. PMID 16234071
- [Background] Mizokami M, Gojobori T, Ohba K, Ikeo K, Ge XM, Ohno T, Orito E, Lau JY. Hepatitis C virus types 7, 8 and 9 should be classified as type 6 subtypes. J Hepatol. 1996 May;24(5):622-4. doi: 10.1016/s0168-8278(96)80149-8. PMID 8773919
- [Background] Nguyen MH, Keeffe EB. Chronic hepatitis C: genotypes 4 to 9. Clin Liver Dis. 2005 Aug;9(3):411-26, vi. doi: 10.1016/j.cld.2005.05.010. PMID 16023974
- [Background] Lu L, Nakano T, He Y, Fu Y, Hagedorn CH, Robertson BH. Hepatitis C virus genotype distribution in China: predominance of closely related subtype 1b isolates and existence of new genotype 6 variants. J Med Virol. 2005 Apr;75(4):538-49. doi: 10.1002/jmv.20307. PMID 15714489
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Lindsay KL. Introduction to therapy of hepatitis C. Hepatology. 2002 Nov;36(5 Suppl 1):S114-20. doi: 10.1053/jhep.2002.36226. PMID 12407584
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Kinzie JL, Naylor PH, Nathani MG, Peleman RR, Ehrinpreis MN, Lybik M, Turner JR, Janisse JJ, Massanari M, Mutchnick MG. African Americans with genotype 1 treated with interferon for chronic hepatitis C have a lower end of treatment response than Caucasians. J Viral Hepat. 2001 Jul;8(4):264-9. doi: 10.1046/j.1365-2893.2001.00292.x. PMID 11454177
- [Background] Muir A, Rockey DC. Treatment of acute hepatitis C with interferon alfa-2b. N Engl J Med. 2002 Apr 4;346(14):1091-2. No abstract available. PMID 11936122
- [Background] Reddy KR, Hoofnagle JH, Tong MJ, Lee WM, Pockros P, Heathcote EJ, Albert D, Joh T. Racial differences in responses to therapy with interferon in chronic hepatitis C. Consensus Interferon Study Group. Hepatology. 1999 Sep;30(3):787-93. doi: 10.1002/hep.510300319. PMID 10462387
- [Background] Wiley TE. Hepatitis C: does race really matter? Am J Gastroenterol. 2001 Aug;96(8):2292-4. doi: 10.1111/j.1572-0241.2001.04030.x. No abstract available. PMID 11513163
- [Background] Hui CK, Yuen MF, Sablon E, Chan AO, Wong BC, Lai CL. Interferon and ribavirin therapy for chronic hepatitis C virus genotype 6: a comparison with genotype 1. J Infect Dis. 2003 Apr 1;187(7):1071-4. doi: 10.1086/368217. Epub 2003 Mar 7. PMID 12660921
- [Background] Dev AT, McCaw R, Sundararajan V, Bowden S, Sievert W. Southeast Asian patients with chronic hepatitis C: the impact of novel genotypes and race on treatment outcome. Hepatology. 2002 Nov;36(5):1259-65. doi: 10.1053/jhep.2002.36781. PMID 12395338
- [Background] McHutchison JG, Gordon SC, Schiff ER, Shiffman ML, Lee WM, Rustgi VK, Goodman ZD, Ling MH, Cort S, Albrecht JK. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. N Engl J Med. 1998 Nov 19;339(21):1485-92. doi: 10.1056/NEJM199811193392101. PMID 9819446